CLINICAL TRIAL: NCT01589289
Title: Rapid Diagnostic Tests in Association With Clinical and Laboratory Predictors for the Diagnosis of Neglected Tropical Diseases in Patients With Neurological Disorders in Rural Hospitals of Bandundu,Democratic Republic of Congo
Brief Title: Rapid Diagnostic Tests and Clinical/Laboratory Predictors of Tropical Diseases in Neurological Disorders in DRC
Acronym: Nidiag-Neuro
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WP2-01-NEU
Record Dates: First submitted 2012-04-26; First posted 2012-05-01 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Neurological Disorders; Cerebral Malaria; Bacterial Meningitis; Central Nervous System Tuberculosis; Neurosyphilis; Cryptococcal Meningitis
Keywords: Diagnostic research; Rapid diagnostic tests; Neurological disorders; Neglected Tropical Diseases; Developing countries
MeSH Terms: conditions — Nervous System Diseases; Malaria, Cerebral; Meningitis, Bacterial; Tuberculosis, Central Nervous System; Neurosyphilis; Meningitis, Cryptococcal; Neglected Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase 3 RDTs (Experimental): The different interventions will be assessed for estimation of sensitivity, specificity and predictive values in the patients' cohort, for the respective target conditions. [To be noted that, in addition, also the predictive values of validated RDTs when used alone and in various combinations will be estimated].
  Interventions: Device: Immunochromatographic HAT tests (DSD); Device: Card Agglutination Trypanosoma Test; Device: TB POC Nucleic Acid Amplification Test (Molbio Diagnostics); Device: TB 3-marker RDT (Tulip diagnostics); Device: Cryptococcal Antigen Lateral Flow Assay (Immy)

INTERVENTIONS:
Device: Immunochromatographic HAT tests (DSD) — Immunochromatographic HAT diagnostic tests manufactured by DSD, Korea and FIND
Device: Card Agglutination Trypanosoma Test — Card Agglutination Trypanosoma Test on whole blood and as dilution
  Other Names: CATT
Device: TB POC Nucleic Acid Amplification Test (Molbio Diagnostics) — TB POC Nucleic Acid Amplification Test: "microPCR handheld device" (Molbio Diagnostics PVT ltd, India)
  Other Names: NAAT
Device: TB 3-marker RDT (Tulip diagnostics) — TB 3-marker RDT: ADA2/IFN-g/LAM (Tulip diagnostics, ltd, India) - pending availability for phase 3 validation
Device: Cryptococcal Antigen Lateral Flow Assay (Immy) — Cryptococcal Antigen Lateral Flow Assay (Immy, USA)
  Other Names: CrAg-LAT

SUMMARY:
The impact of neurological disorders is enormous worldwide, and it is increased in poor settings, due to lack of diagnosis and treatment facilities as well as delayed management. In sub-Saharan Africa, the few observational studies conducted for the past 20 years show that neurological disorders accounted for 7 to 24% of all admissions. Central nervous system (CNS) infections were suspected in one third of all patients admitted with neurological symptoms, with a specific microbial aetiology identified in half of these. Most CNS infections may be considered as "severe and treatable diseases", e.g. human African trypanosomiasis (HAT), cerebral malaria, bacterial meningitis, CNS tuberculosis etc. If left untreated, death or serious sequels occur (mortality rates were as high as 30% in the above mentioned studies), but the outcome may be favourable with timely and appropriate management.

In poor settings, such conditions should be targeted in priority in the clinical decision-making process. Unfortunately, most neuro-infections present with non-specific symptoms in their early stages, leading to important diagnostic delays. Moreover, they require advanced diagnostic technology, which is not available in most tropical rural settings: here, you have to rely on clinical judgment and first-line laboratory results, whose confirming or excluding powers are limited or unknown. Several rapid diagnostic tests (RDTs) have been recently developed for conditions like malaria or HIV, but their diagnostic contribution has not been evaluated within a multi-disease approach.

Thus, this research aims at improving the early diagnosis of severe and treatable neglected and non-neglected infectious diseases which present with neurological symptoms in the province of Bandundu, Democratic Republic of Congo (DRC), by combining classic clinical predictors with a panel of simple point-of-care rapid diagnostic tests.

The evaluation of existing algorithms and elaboration/validation of new guidelines will be described in a subsequent protocol.

DETAILED DESCRIPTION:
The impact of neurological disorders is enormous in terms of mortality, morbidity, physical disability and psychological distress, and it is increased in low-resource settings by lack of diagnosis and of treatment facilities as well as delayed management. The frequency of neurological disorders and the pattern of causative conditions are little documented in low-resource primary care settings.In sub-Saharan Africa, the few observational studies conducted for the past 20 years, show that neurological disorders accounted for 7 to 24% of all admissions. Central nervous system (CNS) infections were suspected in one third of all patients admitted with neurological symptoms, with a specific microbial aetiology identified in half of these. Where it has been investigated, up to one third of neurological admissions was related to HIV infection in some settings. Neuro-infections were also the leading aetiologies of common neurological symptoms (such as headache) in African HIV-positive patients, and autopsy studies have demonstrated that CNS infections accounted for 20% of the causes of death in HIV-positive individuals in sub-Saharan Africa.

Most CNS infections may be considered as "severe and treatable diseases", e.g. human African trypanosomiasis (HAT), cerebral malaria, bacterial meningitis, CNS tuberculosis, neurosyphilis, cryptococcal meningitis or toxoplasma encephalitis etc. If left untreated, death or serious sequels usually occur; mortality rates of neurological admissions were as high as 30% in the above mentioned studies. However, outcome may be favourable with timely and appropriate management.

In resource-constrained settings more than elsewhere, such "severe and treatable" conditions should be targeted in priority in the clinical decision-making process. Unfortunately, most neuro-infections present with non-specific symptoms in their early stages, leading to important diagnostic delays. Moreover, neurological diagnoses frequently require advanced technology, but this is far beyond reach of most tropical rural settings, where you have to rely on clinical judgment and first-line laboratory results. However, the confirming or excluding powers of most clinical and laboratory features are limited or have never been adequately quantified, in particular in settings lacking reference diagnostic methods. Several rapid diagnostic tests (RDTs) have been developed in the last decade for conditions like malaria or HIV infection, but their diagnostic contribution has never been evaluated within a multi-disease approach. Most CNS infections with worldwide distribution affect disproportionally the (sub)-tropical regions, while others are restricted to the tropics. Also, many infections with potential neuropathogenicity belong to the group of 17 Neglected Tropical Diseases (NTDs) on which attention has been recently brought. As said above, most of them may be considered as "severe and treatable"; however, in most tropical settings, epidemiology of NTDs and other infectious diseases (IDs) is largely unknown, seriously impairing the case finding and clinical decision-making.

The aim of this research therefore is to improve the early diagnosis of severe and treatable neglected and non-neglected infectious diseases which may present with neurological symptoms in the province of Bandundu, Democratic Republic of Congo (DRC). This will be achieved through the elaboration and validation of new diagnostic guidelines based on epidemiological evidence, combining classic clinical predictors with a panel of simple point-of-care rapid diagnostic tests, and designed with a "panoramic" (not-to-miss) approach.

In particular, the investigators hope to determine the pre-test probability of HAT and other priority neglected tropical diseases/infectious diseases in patients presenting with neurological disorders; to assess the predictive weight of clinical and first-line laboratory features in the diagnosis of HAT and other priority NTDs/IDs; to assess the sensitivity, specificity and predictive values of novel point-of-care RDTs for the diagnosis of HAT and other priority NTDs/IDs in patients with neurological disorders; and to assess the diagnostic performances of combinations of novel and existing RDTs for diagnosing HAT and other priority NTDs/IDs in patients with neurological disorders. Enrolled patients will be managed according the current standard of care in Bandundu, DRC and with the treatments locally available through health facilities/programs.

The objectives and methodology of this second step of our research (evaluation of existing algorithms and elaboration/validation of new guidelines) will be described in a subsequent protocol. Another similar study (described in another protocol) will be conducted in parallel to explore the aetiologies of prolonged fever in the same setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 5 years-old AND
* Altered state of consciousness (confusion to coma) OR/AND
* Changes of sleep pattern (daytime slumber, night insomnia)OR/AND
* Cognitive decline OR/AND
* Changes in personality/behaviour (e.g. bouts of mania)OR/AND
* Epileptic seizure(s)OR/AND
* Daily severe/progressive headache OR/AND
* Meningismus (headache, neck stiffness, nausea/vomiting, photophobia)
* Cranial nerve lesions OR/AND
* Sensory-motor deficits or other focal neurological signs (e.g. dysphagia, dysarthria, ataxia, dystonia,...)OR/AND
* Gait disorders (e.g. spastic or ataxic gait)

Exclusion Criteria:

* Those unwilling or unable to give written informed consent (either directly or via proxy)
* Those unable in the physician's opinion to comply with the study requirements
* Neurological symptom unequivocally related with recent trauma
* Neurological symptom as sequelae of previous well-established neurological events (e.g. stroke,…)
* First seizure below 6 years of age (early onset seizure)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2012-09; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of HAT and other NTDs/IDs | 18 months
  Number of patients diagnosed with HAT and other NTDs/IDs among those presenting with neurological disorders in rural hospitals of Bandundu, DRC (pre-test probability)
Identification of reliable diagnostic tests | 18 months
  Assessment of the sensitivity, likelihood ratios and performances (diagnostic accuracy) of the novel study RDTs for the respective target conditions, and identification of those that should be included in future diagnostic protocols
Predictive values of RDTs | 18 months
  Predictive values (post-test probabilities) of novel and existing RDTs, alone and in combination, for the respective target conditions within this multi-disease approach
Identification of clinical and laboratory diagnostic indicators | 18 months
  Assessment of the specificity of the different clinical and first-line laboratory features for the diagnosis of HAT and other priority NTDs/IDs in the setting, for determining those that should be included in future diagnostic protocols

SECONDARY OUTCOMES:
Cure rate | 18 months
  Number of patients who positively respond to specific/empirical therapies, as assessed as final patient outcomes (cure, referral, sequelae, death)
Cost-effectiveness of the diagnostic tests | 18 months
  Unit costs of diagnostic tests for the diagnosis of HAT and other priority NTDs/IDs in the setting

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bottieau, MD, Study Director — ITM; Marleen Boelaert, MD, PhD, Study Chair — ITM
Locations (1):
- Reference Hospital Mosango, Mosango, Bandundu, Democratic Republic of the Congo